CLINICAL TRIAL: NCT06080438
Title: The Effect of Topical Botulinum Toxin Eyedrop on Palpebral Fissure Height, Ocular Surface and Tearing
Brief Title: Effect of Topical Botulinum Toxin Eyedrop on Palpebral Fissure
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Patient recruitment shortage and study coordinator turnover
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Wendy Lee, Professor of Clinical, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20220083
Record Dates: First submitted 2023-10-05; First posted 2023-10-12 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Tears; Excess; Eyelid Spasm
MeSH Terms: conditions — Lacerations; Blepharospasm | interventions — Botulinum Toxins; Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Botulinum toxin group (Experimental): The left eye of each participant will receive botulinum toxin eye drops and will remain in this group for up to 40 minutes.
  Interventions: Drug: Botulinum toxin

INTERVENTIONS:
Drug: Botulinum toxin — 15 units of botulinum toxin administered one time to the eye via eye drops
  Other Names: BOTOX

SUMMARY:
The purpose of this research study is to test if Topical (applied to the surface of the eye) Botulinum Toxin temporarily lowers the upper eyelid and makes the eyelid appear less open and thereby affects the eye surface and decreases reflexive tearing.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and above that present to the oculoplastic and reconstructive surgery department that are able to provide informed consent to participate
* Presence of upper eyelid retraction or asymmetry( >1mm)

Exclusion Criteria:

* Adults unable to consent
* Individuals less than 18 years of age
* Prisoners
* Pregnant women. o Patients will be asked if they are pregnant by research staff before participation in the study.

Women who are breast-feeding

* Known contradictions or sensitivities to study medication
* Grossly abnormal lid margins, anatomical abnormalities
* Variable ptosis or eyelid position (e.g., myasthenia gravis, blepharospasm)
* Any ocular or systemic condition that, in the opinion of the investigator, would confound study data, interfere with the subject's study participation, or affected the subject's safety or trial parameters
* Presence of an active ocular infection
* Inability to sit comfortably for 15 - 30 minutes
* Botulinum toxin injection in the eyelids during the past 3 weeks.
* Neuromuscular disorders (e.g., Parkinson's disease or myasthenia gravis)
* Medication use known to interfere with the effects of botulinum toxin-A within the previous 1 month (e.g., aminoglycoside or benzodiazepines),
* Previous history of hypersensitivity reactions to botulinum toxin-A
* Dysfunction of tear production or secretion (e.g., meibomian gland dysfunction or Sjogren's syndrome),

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2024-07-28 (Actual); Study Completion 2024-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Lee, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For interim analysis of futility, the investigators conducted the study with BT eye drops on first 10 patients and then evaluate the results to see if there are any significant effects. If clinically significant effects are seen, then 34 patients totally (17 in BT vs 17 in saline) are included. The study was terminated and did not continue; therefore, only the first phase of the study was conducted with only one arm (BT eye drops) with results reported for the first phase only.
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | Botulinum Toxin Group
Started | 2; 2 eyes
Completed | 0; 0 eyes
Not Completed | 2; 2 eyes
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Units Other Than Participants: eyes
Arm/Group | Botulinum Toxin Group
Number analyzed (Participants) | 2
Number analyzed (eyes) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Palpebral fissure [Mean (Standard Deviation); unit: mm] — Palpebral fissure is the area between the upper and lower eyelid margins. Palpebral fissure height on eyes is measured in primary gaze position with a clear ruler held in a central vertical position between the upper and lower eyelid margin.
  mm | 11.75 (0.42)

OUTCOME MEASURES:

1. Primary Outcome: Change in Palpebral Fissure Height
Description: Palpebral fissure on Day 3 minus palpebral fissure at baseline.
  Palpebral fissure is the area between the upper and lower eyelid margins. Palpebral fissure height on eyes is measured in primary gaze position with a clear ruler held in a central vertical position between the upper and lower eyelid margin.
Time Frame: baseline and Day 3
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: eyes
Arm/Group | Botulinum Toxin Group
Number analyzed (Participants) | 2
Number analyzed (eyes) | 2
mm | -0.5 (0.69)

2. Secondary Outcome: Corneal Staining Density
Description: Scoring of the ocular surface will be done by fluorescein staining and evaluating with a slit lamp and grading scale: 0-3 0 (no punctate staining)
  1. (sparse density)
  2. (moderate density)
  3. (high density and overlapping lesions).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Botulinum Toxin Group
Number analyzed (Participants) | 2
Number analyzed (eyes) | 2
score on a scale | 2 (0)

3. Secondary Outcome: Corneal Staining Density
Description: as for outcome 2
Time Frame: Day 3
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Botulinum Toxin Group
Number analyzed (Participants) | 2
Number analyzed (eyes) | 2
score on a scale | 2 (0)

4. Secondary Outcome: Change in Tearing
Description: Change in tearing will be calculated as tearing on Day 3 minus tearing at baseline.
  Tearing will be assessed using the Schirmer test with anesthesia. Schirmer strip is inserted into the lower conjunctival sac at the junction of the lateral and middle thirds, avoiding touching the cornea, and the length of wetting strips in millimeters is recorded after 5 minutes.
  The result can range from a minimum of 0 mm (no tearing) to a maximum of 35 mm (maximum tearing).
Time Frame: baseline and Day 3
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: eyes
Arm/Group | Botulinum Toxin Group
Number analyzed (Participants) | 2
Number analyzed (eyes) | 2
mm | 3 (5.54)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Botulinum Toxin Group
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
For interim analysis of futility, the investigators conducted the study with BT eye drops on the first 10 patients and then evaluated the results to see if there were any significant effects. If clinically significant effects are seen, then 34 patients totally (17 in BT vs 17 in saline) are included. The study was terminated and did not continue; therefore, only the first phase of the study was conducted with only one arm (BT eye drops) with results reported for the first phase only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/38/NCT06080438/Prot_SAP_000.pdf